CLINICAL TRIAL: NCT04796688
Title: Safety and Efficacy of Universal Chimeric Antigen Receptor-modified AT19 Cells in Patients With CD19+ Relapsed/Refractory Hematological Malignancies: a Single-center, Open-label, Single-arm Clinical Study
Brief Title: Universal Chimeric Antigen Receptor-modified AT19 Cells for CD19+ Relapsed/Refractory Hematological Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Chengdu USino Technology Biology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Proferssor, Cheif Doctor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Universal AT19 cells
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Acute Lymphoblastic Leukemia; Chronic Lymphoblastic Leukemia; B-cell Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Cyclophosphamide + AT19 cells (Experimental): Patients will received lymphodepletion with fludarabine (30 mg/kg) and cyclophosphamide (300 mg/kg) on days -5, -4, and -3, followed by the infusions of AT19 cells on day 0-2. The study will be divided into three groups: B-ALL, B-CLL, and B-cell lymphoma. Doses of 0.5×10^7, 1.0×10^7, and 2.0×10^7 CAR+ T cells (with an allowance of ±20%) will be tested in each group in the 3+3 dose-escalation study. Each dose group has 3 patients. If no DLT emerges in the group, then the next group uses the subsequent higher dose. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level.The maximum dose could be extended.
  Interventions: Drug: Fludarabine + Cyclophosphamide + CAR-NK-CD19 Cells

INTERVENTIONS:
Drug: Fludarabine + Cyclophosphamide + CAR-NK-CD19 Cells — fludarabine 30 mg/kg on day -5, -4, and -3; cyclophosphamide 300 mg/kg on day -5, -4, and -3; CAR-NK-CD19 Cells on day 0.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the primary safety and efficacy of universal chimeric antigen receptor-modified AT19 cells in patients with relapsed or refractory hematological malignancies.

DETAILED DESCRIPTION:
* Adoptive transfer of autologous anti-CD19 CAR-T cells can induce durable remissions in patients with relapsed/refractory hematologic malignancies, including CD19+ B-cell acute lymphoblastic leukemia(B-ALL), B-cell chronic lymphoblastic leukemia(B-CLL), and B-cell lymphoma.
* However, multiple challenges exist for manufacturing CAR-T cells from patients with advanced disease including inability to manufacture a product, disease progression or death while waiting for the CAR-T product to be available, and heterogeneity among autologous CAR-T products that contributes to unpredictable and variable clinical activity.
* Healthy donor T cells can provide a source for production of universal CAR-T cells when combined with gene editing to prevent expression of endogenous TCRs and avoid generation of GvHD in HLA mismatched recipients.
* Cord blood derived T cells from healthy donor are the source for production of universal anti-CD19 CAR-modified AT19 cells. CRISPR/cas9 gene-editing technology has been used to knockout TCRs and HLA-I to avoid GvHD and transplant rejection.
* AT19 cells have exhibited potent cytotoxicity in CD19+ tumor cells and can effectively eradicate CD19+ tumor cells in xenograft mice models, without showing GvHD.
* This study aims to evaluate prelimary safety and efficacy of the universal AT19 cells in patients with relapsed/refractory B-ALL, B-CLL, and B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14-78 years old (including 14 and 78 years old).
2. Clinical diagnosis of CD19+ B-cell hematological malignancies, including acute lymphoblastic leukemia, chronic lymphocytic leukemia and lymphoma.
3. Refractory/Relapsed B-cell malignancies:

   A. Refractory/relapsed B-cell lymphoblastic leukemia, meeting one of the following criteria:

   i. Recurrence within 6 months after first remission. ii. Primary refractory disease which cannot achieve complete remission (CR) after 2 cycles of standardized chemotherapy regimen.

   iii. Failure to achieve CR or relapse after one line or multiple lines of salvage chemotherapy.

   iv. Not suitable for hematopoietic stem cell transplantation (HSCT), or abandon HSCT due to various restrictions, or relapse after HSCT.

   B. Refractory/relapsed B-cell lymphoma, meeting 1 of the first 4 items plus item 5: i. Tumor shrinkage less than 50% or disease progression after 4 cycles of standard chemotherapy.

   ii. Achieved CR after standard chemotherapy, but relapsed within 6 months. iii. 2 or more relapses after CR. iv. Not suitable for HSCT, or abandon HSCT due to various restrictions, or relapse after HSCT.

   v. Subjects must have received adequate treatment in the past, including anti-CD20 monoclonal antibody and combination chemotherapy with anthracyclines.
4. Having a measurable or evaluable lesion:

   A. Patients with lymphoma require a single lesion≥15mm or 2 or more lesions≥10mm.

   B. Patients with leukemia require persistent positive or positive relapse of bone marrow MRD.
5. The toxicity related to previous treatments had returned to < 1 level at enrollment (except for low grade toxicity such as alopecia).
6. Patients have good main organs functions:

   A. Liver function: ALT/AST < 2.5 times the upper limit of normal (ULN) and total bilirubin≤ 1.5 times ULN; B. Renal function: Creatinine clearance rate ≥ 60ml/min. C. Pulmonary function: Indoor oxygen saturation ≥ 95%. D. Cardiac Function: Left ventricular ejection fraction (LVEF) ≥50%, no clinically-significant ECG findings.
7. Estimated survival time≥3 months.
8. Patient or his or her legal guardian voluntarily participates in and signs an informed consent form.

Exclusion Criteria:

1. Central nervous system is involved in leukemia and lymphoma.
2. Known HIV positive patients.
3. CNS diseases, such as epilepsy, cerebral ischemia / hemorrhage, dementia, cerebellar diseases or any CNS related autoimmune diseases.
4. NYHA class III or higher cardiac failure, or with malignant arrhythmia.
5. Myocardial infarction, angioplasty or stent placement, unstable angina or other clinically significant heart history within 12 months before enrollment.
6. Patients who need immediate treatment to control tumor progression or relieve tumor burden.
7. Active autoimmune diseases requiring systemic immunosuppressive therapy.
8. History of symptomatic deep vein thrombosis or pulmonary embolism within 6 months before enrollment.
9. Severe immediate hypersensitivity to any drug to be used in this study.
10. Women who are pregnant or breastfeeding.
11. Other unsuitable conditions in the researchers' opinion.

Ages: 14 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2023-03-10 (Estimated); Study Completion 2024-03-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | within 2 years after infusion
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0).

SECONDARY OUTCOMES:
Overall response rate(ORR) of administering AT19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | within 2 years after infusion
  ORR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Complete response rate(CRR) of administering AT19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | within 2 years after infusion
  CRR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Progress-free survival(PFS) of administering AT19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | 2 years after infusion
  PFS will be assessed from CAR T cell infusion to death or last follow-up (censored).
Duration of Response(DOR) of administering AT19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | 2 years after infusion
  DOR will be assessed from CAR T cell infusion to death or last follow-up (censored).
Overall survival(OS) of administering AT19 cells in Relapsed/Refractory CD19+ B-cell hematological malignancies. | 2 years after infusion
  OS will be assessed from CAR T cell infusion to death or last follow-up (censored).

OTHER OUTCOMES:
In vivo expansion and survival of AT19 cells | 2 years after infusion
  Quantity of AT19 CAR copies in bone marrow and peripheral blood will be determined by using qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No